CLINICAL TRIAL: NCT01126164
Title: Parent Intervention to Reduce Binge Drinking
Acronym: GOALS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Responsible Party: Principal Investigator, Robert Turrisi, Professor of Biobehavioral Health and Prevention Research Center, Penn State University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: R01AA012529 (NIH)
Record Dates: First submitted 2010-05-17; First posted 2010-05-19 (Estimated); Last update posted 2021-03-16 (Actual); Status verified 2021-03

CONDITIONS: Alcohol Consumption
Keywords: parents; peer; basics; college student drinking
MeSH Terms: conditions — Alcohol Drinking; Alcohol Drinking in College

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- parent handbook (Experimental): parent handbook
  Interventions: Behavioral: Parent Handbook and Peer Basics
- peer basics (Experimental): peer delivered basics
  Interventions: Behavioral: Parent Handbook and Peer Basics
- parent handbook and peer basics (Experimental): parent handbook and peer basics
  Interventions: Behavioral: Parent Handbook and Peer Basics

INTERVENTIONS:
Behavioral: Parent Handbook and Peer Basics — Parent and Peer delivered interventions
  Other Names: Parent Handbook; Peer Delivered BASICS

SUMMARY:
Parent and peer interventions to reduce student drinking

DETAILED DESCRIPTION:
Parent and peer interventions to reduce student drinking:

Efficacy;

Mediation:

Moderation

ELIGIBILITY:
Inclusion Criteria:

* varsity athlete in high school

Exclusion Criteria:

* not a varsity athlete in high school

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 800 (Actual)
Dates: Start 2005-09; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
heavy episodic drinking | 6 months post baseline
  typical daily drinking
heavy episodic drinking | 9 months post baseline
  typical daily drinking
heavy episodic peak drinking | 6 months post baseline
  peak number of drinks in one night
heavy episodic peak drinking | 9 months post baseline
  peak number of drinks in one night

SECONDARY OUTCOMES:
drinking consequences | 9 months post baseline
  frequency of blackouts, hangovers, vomiting, fights, unplanned sex, trouble with police, poor academic performance as measured by the rapi; yaapst (standard instruments used in all college alcohol prevention trials)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Turrisi, Ph.D., Principal Investigator — Penn State University
Locations (1):
- Penn State University, University Park, Pennsylvania, United States

REFERENCES:
- [Result] Turrisi R, Larimer ME, Mallett KA, Kilmer JR, Ray AE, Mastroleo NR, Geisner IM, Grossbard J, Tollison S, Lostutter TW, Montoya H. A randomized clinical trial evaluating a combined alcohol intervention for high-risk college students. J Stud Alcohol Drugs. 2009 Jul;70(4):555-67. doi: 10.15288/jsad.2009.70.555. PMID 19515296